CLINICAL TRIAL: NCT07153718
Title: Optimal Ablation Strategies for Persistent Atrial Fibrillation With Heart Failure - Optimization of Intervention Strategies for Persistent Atrial Fibrillation
Brief Title: Optimal Ablation Strategies for Persistent AF With HF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Xu Liu (Other)
Responsible Party: Sponsor-Investigator, Xu Liu, Dr, Shanghai Chest Hospital
Organization: Shanghai Chest Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXT- AF&HF
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Heart Failure; Persistent Atrial Fibrillation
Keywords: ablation strategy for persistent atrial fibrillation with heart failure
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anatomical-guided Ablation Group (Active Comparator): Patients in the ANAT group would receive anatomical-guided ablation after PVI, including linear ablation and Vein of Marshall (VOM) ethanol infusion.
  Interventions: Procedure: Anatomical-guided Ablation
- Electrogram-guided Ablation Group (Active Comparator): Patients in the EGM group received target electrogram ablation after PVI while did not receive anatomical-guided ablation. We defined the target electrograms into 4 types as follows.(1) Spatial-temporal Dispersion Activation (2) Locally Short Cycle Length Activity (3) High-Frequency Potentials (4) Focal Activity
  Interventions: Procedure: Electrogram-guided ablation
- Extensive Electrogram-Anatomical Guided Ablation Group (Experimental): Patients in the extensive ablation group (EXT group) would receive EGM-guided ablation firstly. The anatomical-guided ablation would be performed after EGM-guided ablation no matter whether AF terminated during EGM-guided ablation.
  Interventions: Procedure: Extensive electrogram-anatomical guided ablation

INTERVENTIONS:
Procedure: Electrogram-guided ablation — pulmonary vein ioslation; target electrograms ablation, including (1) Spatial-temporal Dispersion Activation, (2) Locally Short Cycle Length Activity, (3) High-Frequency Potentials, (4) Focal Activity.
  Arms: Electrogram-guided Ablation Group
Procedure: Anatomical-guided Ablation — pulmonary vein isolation; LA roof, posterior inferior wall and mitral isthmus linear lesion; Vein of Marshall (VOM) ethanol infusion.
  Arms: Anatomical-guided Ablation Group
Procedure: Extensive electrogram-anatomical guided ablation — pulmonary vein isolation; target electrogram ablation; linear ablation
  Arms: Extensive Electrogram-Anatomical Guided Ablation Group

SUMMARY:
Atrial fibrillation (AF) in the context of heart failure (HF) is associated with a markedly poor prognosis. Catheter ablation has been shown to improve outcomes in this population, enhancing ablation success rates in these patients is critical for further reducing morbidity and mortality. We conducted this multicenter, randomized clinical trial to systematically evaluate the optimal ablation strategy in patients with heart failure and persistent AF.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) in the context of heart failure (HF) is associated with a markedly poor prognosis, with one-year all-cause mortality rates approaching 34% and substantially elevated risks of stroke and rehospitalization. Catheter ablation has been shown to improve outcomes in this population, as evidenced by numerous pivotal studies, such as CASTLE-AF. It is well recognized that the majority of patients with HF and AF exhibit persistent AF; however, the underlying mechanisms responsible for sustaining persistent AF in this population remain to be fully elucidated. Thus, enhancing ablation success rates in these patients is therefore critical for further reducing morbidity and mortality.

Building on prior research, we have identified driver regions as critical determinants in the maintenance of persistent atrial fibrillation. Moreover, our randomized controlled trials have demonstrated that electro-anatomical ablation may represent the optimal strategy for persistent AF. Based on these findings, we conducted a multicenter, randomized clinical trial to systematically evaluate the optimal ablation strategy in patients with heart failure and persistent AF.

ELIGIBILITY:
Inclusion Criteria:

* All inclusion criteria must be met to be included in the study.

  1. Age: Patients aged 18-80 years, with persistent atrial fibrillation (AF) and heart failure (HF), regardless of ejection fraction (EF).
  2. Diagnosis of Heart Failure:

     Heart Failure with Reduced Ejection Fraction (HFrEF): LVEF ≤ 40%. Heart Failure with Preserved Ejection Fraction (HFpEF): LVEF > 40%, including HFmrEF (LVEF 41-50%).
  3. Symptomatic Atrial Fibrillation: Patients with symptomatic persistent AF who have failed or are intolerant to at least one antiarrhythmic drug.
  4. NYHA Class II-III: Patients with heart failure classified as NYHA class II-III, who are symptomatic despite optimal medical therapy. Informed Consent: Able to provide written informed consent for participation in the study.
  5. Guideline-Recommended Pharmacologic Therapy: Patients who have received and are currently on guideline-recommended pharmacologic therapy for heart failure, including but not limited to ACE inhibitors, beta-blockers, diuretics, and mineralocorticoid receptor antagonists (MRAs).

Exclusion Criteria:

* Any of the following criteria shall be excluded.

  1. End-Stage Heart Failure: Patients with heart failure classified as NYHA class IV or with LVEF ≤ 20%.
  2. Severe Comorbidities:
  3. Patients with severe pulmonary disease (e.g., COPD, severe restrictive lung disease).
  4. Severe renal dysfunction (eGFR < 30 mL/min/1.73m²) or advanced liver disease.
  5. Active malignancy or other terminal illnesses with a prognosis of less than one year.
  6. Inability to Tolerate Ablation:

  <!-- -->

  1. Patients unable to undergo catheter ablation due to anatomical or procedural issues.
  2. Patients with contraindications to the procedure, including allergy to contrast agents or inability to tolerate anesthesia.
  3. Left atrial thrombus confirmed by preoperative esophageal ultrasound; 7. Uncontrolled Arrhythmias: Patients with persistent or paroxysmal AF who are unable to maintain sinus rhythm despite optimal medical therapy or require frequent hospitalization for arrhythmia control.

  8. Pregnancy: Pregnant or breastfeeding women. 9. Contraindications to Anticoagulation: 10. Patients who are contraindicated for anticoagulation therapy (e.g., history of major bleeding or bleeding diathesis).

  11. History of Severe Valve Disease: Patients with a history of severe valve disease and/or prosthetic valve replacement.

  12. Recent Myocardial Infarction or Stroke: Patients who have had a myocardial infarction or stroke within the past 3 months.

  13. Contrast Agent Allergy: Patients with a known allergy to contrast agents. 14. Contraindications for Cardiac Catheterization: Any contraindications for cardiac catheterization, including inability to safely perform the procedure.

  15. Atrial Fibrillation Ablation: Patients who have previously undergone atrial fibrillation ablation.

  16. Cardiac Surgery: Patients who have undergone any cardiac surgery within the last 2 months.

  17. Life Expectancy: Patients with a life expectancy of less than 1 year.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
a composite of cardiovascular mortality, hospitalization or urgent visits | 12, 18, 24, 36, 46, 60months
  The primary endpoint was the incidence of a composite of cardiovascular mortality, hospitalization or urgent visits due to worsening heart failure during the follow-up period after a single catheter ablation procedure
freedom from any documented AF/AT | 12, 18, 24, 36, 48, 60months
  freedom from any documented AF/AT episode lasting more than 30 seconds after the blanking period without anti-arrhythmic drug treatment

SECONDARY OUTCOMES:
AF burden <1% | 12, 24, 36, 48, 60 months after a single procedure
  AF burden <1% after a single ablation procedure, as measured by Holter monitoring or device-recorded data (Patients who remained in persistent AF throughout follow-up were assigned AF burden=100%. Both ends of the distribution (burden=0% and burden=100%) were included in statistical analysis.).
Improvement in New York Heart Association (NYHA) functional class | 12, 24, 36, 48, 60 months after a single procedure
  Improvement in New York Heart Association (NYHA) functional class by at least one grade
Change in 6-minute walk test | 12, 24, 36, 48, 60 months after a single procedure
  Change in 6-minute walk test from baseline to Month 3, 12, 24, 36, 48, 60 months after a single procedure
Change in N-terminal pro-B type natriuretic peptide (NT-proBNP) | Month 3,12, 24, 36, 48, 60 after a single procedure
  Change in N-terminal pro-B type natriuretic peptide (NT-proBNP) from baseline to Month 3,12, 24, 36, 48, 60 after a single procedure
Incidence of procedure-related complications | 30 days after a single procedure
  Incidence of procedure-related complications, including but not limited to: vascular complications (e.g., hematoma, pseudoaneurysm), cardiac tamponade, stroke or transient ischemic attack (TIA), phrenic nerve injury, atrioesophageal fistula, procedure-related death within 30 days.

CONTACTS AND LOCATIONS:
Locations (10):
- China (10):
  - The PLA Navy Anqing Hospital, Anqing, Anhui
  - The Central Hospital of Wuhan, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Changshu Hospital of Traditional Chinese Medicine, Changshu, Jiangsu
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Second Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong
  - Jinan City People's Hospital, Jinan, Shandong
  - Affiliated Hospital of Jining Medical University, Jining, Shandong
  - Yuhuan Second People's Hospital, Yuhuan, Zhejiang
  - Shanghai Jiao Tong University School of Medicine, Shanghai Chest Hospital, Shanghai
  - Ren Ji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) from this study will not be shared publicly due to concerns regarding patient confidentiality and the sensitive nature of medical data. Given the potential risks of identifying participants from detailed clinical information, the data will remain confidential and will not be made available for public sharing. Additionally, the study involves proprietary methodologies and ongoing analyses that are part of the intellectual property of the institution. As such, sharing the IPD at this stage could compromise the integrity of the study's findings and its future applications.